CLINICAL TRIAL: NCT06724107
Title: Effect of Photofunctionalization With on Titanium Dental Implants. A Pilot Sutdy
Brief Title: Photofunctionalization With UVC
Acronym: EPID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate Profesor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.I. 23/523-EC_P
Record Dates: First submitted 2023-09-22; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Implant Site Reaction
Keywords: ISQ (implant stability quotient); inmediate loading; UVC; dental implants

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UVC group (Experimental): photofunctionalised (study group) implants
  Interventions: Radiation: UVC
- Control group (Placebo Comparator): non-photofunctionalised (control group) implants
  Interventions: Radiation: UVC

INTERVENTIONS:
Radiation: UVC — It is proposed to evaluate and compare the ISQ at 1 week, 2 weeks, 3 weeks and 4 weeks in patients undergoing implant placement surgery by comparing photofunctionalised (study group) and non-photofunctionalised (control group) implants in both native bone and grafted bone. To assess whether immediate loading can be carried out before 4 weeks and how long the waiting time for implant loading can be reduced, by performing predictability curves.

SUMMARY:
Summary:

Objective: The general objective is to compare the placement of standard implants with a surface photofunctionalization technique based on ultraviolet C radiation (UVC), having as working hypothesis that this photofunctionalization will accelerate the bone apposition on the implant surface and increase the amount of bone that binds to the implant, making it possible to load these photofunctionalized implants in less time.

Design: Pilot, clinical, randomized, prospective, controlled, single-center, prospective study.

Scope of the study: Master's Degree in Oral Surgery and Implantology. Faculty of Dentistry. Complutense University of Madrid.

Subjects of the study: patients attending the Master's Degree in Oral Surgery and Implantology for rehabilitation with dental implants, regardless of the sector in which they have missing teeth.

Key words: ISQ (implant stability quotient), inmediate loading, UVC, dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients requiring dental implant surgery with or without bone or soft tissue regeneration surgery.
* Acceptance of the informed consent document.

Exclusion Criteria:

* Subjects with systemic diseases leading to untreated or uncontrolled haemostasis or coagulation disturbances.
* Subjects with active infectious diseases (tuberculosis, HIV, syphilis, hepatitis, etc).
* Patients under pharmacological treatment with monoclonal antibodies, bisphosphonates, chemotherapy or prolonged treatment with corticoids.
* Patients with alcoholism or drug addiction.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-12 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Bone regeneration | 3 months
  Bone implant contact (BIC) Histotogic parameter in percentage

SECONDARY OUTCOMES:
ISQ and marginal bone loss | 12 months
  Implant stability quotient and marginal bone loss measure with X-rays (quantitative parameter)

CONTACTS AND LOCATIONS:
Overall Officials: isabel leco, PhD, Study Director — UCM
Locations (1):
- Jesus Torres, Madrid, Spain